CLINICAL TRIAL: NCT05195489
Title: Examining the Impact of Family Connectors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-01486; P50MH113662 (NIH)
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Caregiver Stress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Intervention (Experimental): Family members participate in Connectors by phone and receive a packet of resources
  Interventions: Other: Family Connectors
- Comparison (No Intervention): Family members receive a pack of resources

INTERVENTIONS:
Other: Family Connectors — The Family Connectors Program is a manualized program that uses a time-limited parent-to parent (i.e. peer parent) support and education program delivered by phone to families of youth with serious mental health difficulties, assisting family members in becoming fully engaged with provider teams who coordinate and provide care. Family Connectors is delivered weekly by phone over the course of between three and six months.
  Arms: Active Intervention

SUMMARY:
The purpose of this study is to understand the impact of Family Connectors, a peer-to-peer support and education program for family members who have participated in OnTrackNY, a treatment program for adolescents and young adults.

DETAILED DESCRIPTION:
The study objectives are to examine the association between involvement in Family Connectors, a manualized peer-to-peer support and education program for family members of adolescents or young adults with symptoms of first episode psychosis, and feelings of empowerment, self-efficacy and social support.

ELIGIBILITY:
Inclusion Criteria:

* English speaking, due to the study materials not being validated in other languages.
* 18 years of age or older,
* Family member of adolescents/young adults with first episode psychosis who participated in OnTrackNY.

Exclusion Criteria:

* Does not provide informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Hoagwood, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Researchers who provide a methodologically sound proposal.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Intervention | Comparison
Started | 11 | 17
Completed | 9 | 13
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Removed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Intervention | Comparison | Total
Number analyzed (Participants) | 9 | 13 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.78 (13.99) | 57.38 (11.84) | 57.95 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 7 | 10 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 3 | 7 | 10
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Perceived Social Support
Description: Perceived social support is measured by a 13-item self-reported questionnaire. The subject is asked to rate each statement about social support on a scale of 1-7 (1=very strongly disagree, 2=strongly disagree, 3=disagree, 4=neither agree nor disagree, 5=agree, 6=strongly agree, 7=very strongly agree). Scores range from 13-91. Higher scores indicate stronger social support.
Time Frame: Month 1, Month 7
Population: The measure was not completed in full by two participants in the comparison group and one participant in the FC group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Intervention | Comparison
Number analyzed (Participants) | 8 | 11
units on a scale | -5.06 (7.39) | 2.91 (8.18)

2. Primary Outcome: Change in Caregiver Strain
Description: Caregiver strain is measured by a 10-tiem self-reported questionnaire. The subject is asked to rate each statement relating to caregiver strain on a scale of 1-5 (1=not at all, 2=a little, 3=somewhat, 4=Quite a bit, 5=very much). Scores range from 10-50, with higher scores indicating high caregiver strain.
Time Frame: Month 1, Month 7
Population: The measure was not completed in full by four participants in the comparison group and one participant in the FC group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Intervention | Comparison
Number analyzed (Participants) | 8 | 9
units on a scale | -2.19 (11.32) | 0.22 (4.41)

3. Primary Outcome: Change in Perceived Self-efficacy
Description: Perceived self-efficacy is measured by a 7-tiem self-reported questionnaire. The subject is asked to rate each statement on a scale of 1-5 (1=strongly disagree, 2=disagree, 3=neither agree nor disagree, 4=agree, 5=strongly agree). Scores range from 7-35, with higher scores indicating greater perceived self-efficacy.
Time Frame: Month 1, Month 7
Population: The measure was not completed in full by one participant in the comparison group and two participants in the FC group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Intervention | Comparison
Number analyzed (Participants) | 7 | 12
units on a scale | -0.29 (3.31) | -0.46 (2.25)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Active Intervention | Comparison
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/17
Other Adverse Events (participants affected / at risk) | 0/11 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT05195489/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT05195489/ICF_000.pdf